CLINICAL TRIAL: NCT00001814
Title: Genetic Analysis of Inherited Urologic Malignant Disorders: Collection of Samples
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990101; 99-C-0101
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-02

CONDITIONS: Neoplastic Syndromes, Hereditary; Urologic Neoplasms
Keywords: Hereditary; Kidney; MET; Oncocytoma; VHL
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary; Urologic Neoplasms; Adenoma, Oxyphilic

SUMMARY:
Investigation of the causes of genetic defects relating to hereditary urologic malignancies will be undertaken. These rare disorders result from inherited or newly arising mutations in genes involved in the development and function of different organ systems. As specific disease syndromes are recognized and the responsible genes identified, mutations in individual families can be identified. Correlation of mutation sites with clinical information will help determine how specific gene segments encode important functional protein domains.

Families with urologic malignant disorders of known or suspected genetic basis will be enrolled. Genetic linkage studies will include all available family members, while gene sequence analysis will be performed on affected individuals. Unaffected family members or unrelated normal individuals will serve as controls. The family members will be identified by the proband or proband's parent when the initial pedigree is taken. Subjects considered by the investigators to be appropriate for linkage studies will be invited to participate by the local genetics provider or by the investigators, who will then connect these members to their own local providers for enrollment.

In our studies of inherited urologic malignant disorders, there may be individuals from renal cancer families who do not undergo clinical evaluation for the presence of an inherited urologic malignant disorder at the National Institutes of Health because of their health problems, geographical location, or personal preference. Even though these individuals do not undergo a clinical evaluation of their suspected inherited urologic malignant disorder at the National Institutes of Health, they may have rare diseases that are extremely important to study. Therefore, we intend to collect blood samples for genetic studies from these individuals to facilitate linkage analysis and disease gene identification. Samples will be collected either by the individual's physician and sent to NIH, or will be collected by NIH physicians at either the individual's off-site location or at the NIH.

DETAILED DESCRIPTION:
Investigation of the causes of genetic defects relating to hereditary urologic malignancies will be undertaken. These rare disorders result from inherited or newly arising mutations in genes involved in the development and function of different organ systems. As specific disease syndromes are recognized and the responsible genes identified, mutations in individual families can be identified. Correlation of mutation sites with clinical information will help determine how specific gene segments encode important functional protein domains.

Families with urologic malignant disorders of known or suspected genetic basis will be enrolled. Genetic linkage studies will include all available family members, while gene sequence analysis will be performed on affected individuals. Unaffected family members or unrelated normal individuals will serve as controls. The family members will be identified by the proband or proband's parent when the initial pedigree is taken. Subjects considered by the investigators to be appropriate for linkage studies will be invited to participate by the local genetics provider or by the investigators, who will then connect these members to their own local providers for enrollment.

In our studies of inherited urologic malignant disorders, there may be individuals from renal cancer families who do not undergo clinical evaluation for the presence of an inherited urologic malignant disorder at the National Institutes of Health because of their health problems, geographical location, or personal preference. Even though these individuals do not undergo a clinical evaluation of their suspected inherited urologic malignant disorder at the National Institutes of Health, they may have rare diseases that are extremely important to study. Therefore, we intend to collect blood samples for genetic studies from these individuals to facilitate linkage analysis and disease gene identification. Samples will be collected either by the individual's physician and sent to NIH, or will be collected by NIH physicians at either the individual's off-site location or at the NIH.

ELIGIBILITY:
Category I: Individuals and family members with established diagnoses of hereditary malignancies where the disease gene is known, specifically von Hippel Lindau or HPRC.

Category II: Individuals and family members with malignant disorders where the disease gene is not yet known, specifically hereditary forms of Type II papillary renal cancer, clear cell renal carcinoma, renal oncocytoma or chromophobe renal carcinoma or Birt Hogg Dube syndrome.

Category III: Malignant diseases of suspected, but not proven genetic etiology, including families with more than one individual affected by the same or related cancers.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 1999-04; Study Completion 2001-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Puck JM, Nussbaum RL, Conley ME. Carrier detection in X-linked severe combined immunodeficiency based on patterns of X chromosome inactivation. J Clin Invest. 1987 May;79(5):1395-400. doi: 10.1172/JCI112967. PMID 2883199
- [Background] Conley ME, Lavoie A, Briggs C, Brown P, Guerra C, Puck JM. Nonrandom X chromosome inactivation in B cells from carriers of X chromosome-linked severe combined immunodeficiency. Proc Natl Acad Sci U S A. 1988 May;85(9):3090-4. doi: 10.1073/pnas.85.9.3090. PMID 2896355
- [Background] Conley ME, Puck JM. Carrier detection in typical and atypical X-linked agammaglobulinemia. J Pediatr. 1988 May;112(5):688-94. doi: 10.1016/s0022-3476(88)80683-8. PMID 2896233